CLINICAL TRIAL: NCT04694404
Title: The Efficacy and Safety of S-1 Plus Oxaliplatin in First-line Treatment of Ederly Patients With Advanced or Recurrent Gastric Cancer
Brief Title: Efficacy and Safety of S-1 Plus Oxaliplatin in First-line Treatment of Ederly Patients With Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aiping Zhou (Unknown)
Responsible Party: Sponsor-Investigator, Aiping Zhou, Chief physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-PI-105
Record Dates: First submitted 2017-11-05; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: S-1 Plus Oxaliplatin
Keywords: S-1,Oxaliplatin,Advanced or Recurrent Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: Single Group Assignment Eledrly Patients with Untreated Advanced or Recurrent Gastric Cancer
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- S-1 Plus Oxaliplatin (Experimental): Oxaliplatin 85 mg/m2 (D1, q2w) and S-1 (40mg BID for body surface area < 1.25 m2; 50mg BID for body surface area of 1.25-1.5 m2; and 60mg BID for body surface area >1.5 m2; D1-10, q2w)
  Interventions: Drug: S-1,Oxaliplatin

INTERVENTIONS:
Drug: S-1,Oxaliplatin — Oxaliplatin 85 mg/m2 (D1, q2w) and S-1 (40mg BID for body surface area < 1.25 m2; 50mg BID for body surface area of 1.25-1.5 m2; and 60mg BID for body surface area >1.5 m2; D1-10, q2w)

SUMMARY:
Elderly patients have poor tolerance and physical condition, we will prove 2-week schedule of oxaliplatin plus S-1 have a good efficacy and a better safety for elderly patients with advanced or recurrent gastric cancer.

DETAILED DESCRIPTION:
3-week plan of S-1 plus Oxaliplatin has been widely used,but it also has cumulative toxicity.Meanwhile elderly patients have poor tolerance and physical condition, we will prove 2-weeks schedule of oxaliplatin plus S-1 have a good efficacy and a better safety for elderly patients with advanced or recurrent gastric cancer.Untreated elderly patients with advanced or recurrent gastric cancer will receive Oxaliplatin 85 mg/m2 (D1, q2w) and S-1(40mg BID for body surface area < 1.25 m2; 50mg BID for body surface area of 1.25-1.5m2; and 60mg BID for body surface area >1.5 m2; D1-10, q2w) as the first-line treatment. We will investigate the efficacy and safety of the combination treatment, and expect to provide a good effective treatment plan and a better safety for elderly patients with advanced or recurrent gastric cancer in China.The primary endpoint is progression-free survival(PFS), and the secondary endpoints are objective response rate(ORR), overall survival(OS) and the safety.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed unresectable or recurrent gastric or gastroesophageal junction adenocarcinoma;
* Aged≥60
* ability of oral administration;
* CT or MRI can be used to assess measurable or non-measurable lesions according to the criteria of Response Evaluation Criteria In Solid Tumours (RECIST 1.1);
* Untreated
* more than 12 months after the last adjuvant/neoadjuvant chemotherapy;
* ECOG=0-2;
* Available organ function: ALT≤2.5xULN;AST≤2.5xULN;If patients have hepaticmetastasis,ALT≤2.5xULN,AST≤2.5xULN;ALP≤2xULN;TBIL≤1.0xULN;NEUT≥1.5×109/L;PLT≥100×109/L;Hb≥90g/L;Creatinine≤1.0xULN;Creatinine Clearance≥60ml/min
* Informed consent;
* Expected survival more than 3 months;More than 3 weeks after major surgery.

Exclusion Criteria:

* Neoadjuvant and/or adjuvant have been treated with more than two plans;
* In the past two years, the total dose of oxaliplatin≥800mg/m2;
* Other cancers in the past 5 years,except for cervical carcinoma in situ or non-melanoma skin cancer;
* Symptomatic brain metastases or soft meningeal metastasis;
* Myocardial infarction (in the last 6 months), severe instability angina, congestive heart failure;
* Serious complications (including intestinal paralysis, gastrointestinal obstruction, interstitial pneumonia, pulmonary fibrosis, uncontrolled diabetes, renal insufficiency and cirrhosis); Chronic nausea, vomiting or diarrhea (more than 4 times per day, or watery);Gastrointestinal bleeding requires regular blood transfusion;HIV or AIDS; Mental illness; Neuropathy grade≥2;Infectious diseases or inflammation, temperature≥38℃;
* Known allergy to drugs in the study;
* Pregnant or lactating women;
* Both male and female subjects of potential fertility have to agree effective birth control during the entire study;
* Experimental drugs used no more than 4 weeks;
* Other conditions the researchers considered ineligible for the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-05-11 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 6 months
  Progression-free survival

SECONDARY OUTCOMES:
ORR | 6 months
  Objective response rate
OS | 1 year
  Overall survival
The number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 1 year
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: Aiping Zhou, Doctor, Study Director — Chinese Academy of Medical Sciences
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese ACademy of Medical Sciences and Peking Union Medical College, Beijing, China

REFERENCES:
- [Derived] Jiang Z, Zhou A, Sun Y, Zhang W. Biweekly oxaliplatin plus S1 for Chinese elderly patients with advanced gastric or gastroesophageal junction cancer as the first-line therapy: a single-arm, phase 2 study. BMC Cancer. 2022 Mar 9;22(1):253. doi: 10.1186/s12885-022-09332-7. PMID 35264150